CLINICAL TRIAL: NCT06515132
Title: Efficacy and Safety of Spinal Cord Stimulation in Patients With Disorders of Consciousness: A Multicenter, Double-blind, Randomized Controlled Trail
Brief Title: Efficacy and Safety of Spinal Cord Stimulation in Patients With Spinal Cord Stimulation
Acronym: SCORS-DOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xuehai Wu, Deputy Director of Shanghai Neurosurgical Emergency Center, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2024-752
Record Dates: First submitted 2024-06-23; First posted 2024-07-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Disorder of Consciousness; Spinal Cord Stimulation
Keywords: Disorder of Consciousness; Spinal Cord Stimulation; Randomized clinical trail
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is being conducted as a double-blind trial, wherein the surgeons, assessors and participants' family members are kept unaware of the assigned research groups. However, it is necessary to inform the physicians responsible for adjustment of stimulation parameters about the allocation of participants. Follow-up assessments of participants after stimulation will be conducted by an independent assessor using standardized evaluation criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCS group (Experimental): SCS stimulation therapy is initiated 1 week post-surgery, which is administered continuously for a duration of 6 months.
  Interventions: Procedure: SCS Stimulation
- Sham group (Sham Comparator): Sham stimulation therapy is initiated 1 week post-surgery, and SCS stimulation therapy is initiated 3 months post-surgery, which is stimulated continuously for a duration of 3 months.
  Interventions: Procedure: Sham Stimulation

INTERVENTIONS:
Procedure: SCS Stimulation — Participants will accept the SCS stimulus for six months
  Arms: SCS group
Procedure: Sham Stimulation — Sham stimulation will be performed in the first three months after surgery, and SCS stimulation will be started in the fourth month after surgery
  Arms: Sham group

SUMMARY:
Investigating the efficacy and safety of spinal cord stimulation for patients with disorders of consciousness.

DETAILED DESCRIPTION:
Disorder of Consciousness (DOC) is a highly significant and concerning consequence that frequently ensues various acute brain injuries. The DOC encompasses coma, unresponsive wakefulness syndrome (UWS), also known as persistent vegetative state (PVS), and minimally conscious state (MCS). Currently, the available treatments for arousing patients with DOC are relatively limited, encompassing pharmacotherapy, hyperbaric oxygen therapy, neuromodulation, physical rehabilitation exercises, and traditional Chinese acupuncture. Among these approaches, only amantadine and transcranial direct current stimulation have demonstrated efficacy in DOC patients; however, further extensive validation is still warranted.

In recent years, spinal cord stimulation (SCS) has emerged as a cutting-edge and extensively researched modality for arousal therapy. SCS is a form of neuromodulation therapy primarily utilized for intractable pain, diabetic neuropathy, and muscle spasticity, the therapeutic efficacy of the SCS is both significant and safe. Although preliminary studies have demonstrated the potential of SCS in promoting arousal in patients with DOC, these findings are currently limited to small sample reports. Therefore, this multicenter randomized controlled trial aims to provide robust evidence on the effectiveness of SCS in promoting arousal among patients with DOC, thereby standardizing its clinical application and offering advanced evidence-based medicine for DOC management.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65, experiencing DOC for a duration ranging from 3 months to 1 year following brain disease.
* Patients diagnosed with DOC as a consequence of traumatic brain injury, hypertensive intracerebral hemorrhage, or severe cerebral infarction.
* Patients exhibiting stable cerebral anatomy and no need for further cranioplasty or hydrocephalus shunt.
* Patients in MCS, who fulfill at least one of the following criteria: ① Demonstrating an oriented response to noxious stimuli; ② Exhibiting sustained eye tracking behavior; ③ Displaying purposeful movements; ④ Manifesting comprehension of language or emotions and actions (often observed in specific environments such as when hearing family members crying).
* The vital signs and state of consciousness are stable: normal body temperature, the spontaneous breathing is stable (minimal sputum production and respiratory stability without oxygen supplementation for at least 2 hours); there is no significant change in the level of consciousness for at least 1 month and more.
* Presence of short-latency responses (N20/P25) on somatosensory evoked potentials (SEP) recorded from the median nerve in the upper limbs.
* Written informed consent obtained from legal guardians or representatives.

Exclusion Criteria:

* Patients with a history of severe neurological or psychiatric disorders, or other significant diseases impacting prognosis prior to the onset of DOC;
* Patients with contraindications for surgery, such as acute infections or coagulation disorders;
* Patients who require short-wave diathermy treatment and are unable to undergo neurostimulation;
* Patients with hypoxic brain injury due to suffocation, cardiac arrest, or respiratory arrest;
* Patients with brainstem hemorrhage;
* Pregnant women;
* Patients who voluntarily request SCS implantation but are unwilling to cooperate with the research protocol;
* Participants in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Effective rate of awakening | SCS stimulation for 3 months after operation
  The CRS-R is employed, with a minimum of 5 CRS-R assessments conducted at each follow-up time point, accompanied by simultaneous video recording. And the highest value is scored as a state of consciousness. The clinical assessment of participants' consciousness is deemed significantly improved when it fulfills the following criteria: a) MCS- recover to consciousness level of MCS+ or higher; b) MCS status (MCS- or MCS+) recover to emergence from MCS (restoration of functional communication).

SECONDARY OUTCOMES:
The difference of CRS-R scale relative to baseline between SCS group and Sham group | SCS stimulation for 14 days, 1-month-postoperative-stimulation, 3-month-postoperative-stimulation, 6-month-postoperative-stimulation
  The Coma Recovery Scale-Revised (CRS-R) is a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness. It has good validity, reliability and practicability.
The difference of SECONDs scale relative to baseline between SCS group and Sham group | SCS stimulation for 14 days, 1-month-postoperative-stimulation, 3-month-postoperative-stimulation, 6-month-postoperative-stimulation
  The Simplified Evaluation of CONsciousness Disorders (SECONDs) is a fast tool to assess consciousness in brain-injured patients.
The difference of modified Ashworth scale relative to baseline between SCS group and Sham group | SCS stimulation for 14 days, 1-month-postoperative-stimulation, 3-month-postoperative-stimulation, 6-month-postoperative-stimulation
  The modified Ashworth scale is the most universally accepted clinical tool used to measure the increase of muscle tone.
The NCS-R scale relative to baseline between SCS group and Sham group | SCS stimulation for 14 days, 1-month-postoperative-stimulation, 3-month-postoperative-stimulation, 6-month-postoperative-stimulation
  The Nociception Coma Scale-Revised (NCS-R) was developed to help assess pain in patients with disorders of consciousness (DOC). Several studies have shown its sensitivity in assessing response to acute noxious stimuli.
The difference of effective rate of awakening between SCS group and Sham group by SECONDs scale | SCS stimulation for 3-month-postoperative-stimulation
SCS stimulation for 6-month-postoperative-stimulation, the difference of effective rate of awakening between SCS group and Sham group by CRS-R scale | SCS stimulation for 6-month-postoperative-stimulation
The difference of effective rate of awakening between SCS group and Sham group by SECONDs scale | SCS stimulation for 6-month-postoperative-stimulation
The difference of recovery trajectories of consciousness level between SCS group and Sham group | SCS stimulation for 6-month-postoperative-stimulation
The difference of effective rate of awakening of 3 month s of sham stimulation and 3 month s of SCS stimulation in Sham group | 6-month-postoperation

OTHER OUTCOMES:
Security outcome | 3 months after operation
  Incidence of postoperative infections within 3 months after operation
Security outcome | 3 months after operation
  Incidence of postoperative hemorrhage within 3 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Xuehai Wu, Ph.D., Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Xiangya Hospital,Central South University, Changsha, Hunan
  - Department of Neurosurgery, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Erp WS, Lavrijsen JC, Vos PE, Bor H, Laureys S, Koopmans RT. The vegetative state: prevalence, misdiagnosis, and treatment limitations. J Am Med Dir Assoc. 2015 Jan;16(1):85.e9-85.e14. doi: 10.1016/j.jamda.2014.10.014. PMID 25528282
- [Background] Maas AIR, Menon DK, Manley GT, Abrams M, Akerlund C, Andelic N, Aries M, Bashford T, Bell MJ, Bodien YG, Brett BL, Buki A, Chesnut RM, Citerio G, Clark D, Clasby B, Cooper DJ, Czeiter E, Czosnyka M, Dams-O'Connor K, De Keyser V, Diaz-Arrastia R, Ercole A, van Essen TA, Falvey E, Ferguson AR, Figaji A, Fitzgerald M, Foreman B, Gantner D, Gao G, Giacino J, Gravesteijn B, Guiza F, Gupta D, Gurnell M, Haagsma JA, Hammond FM, Hawryluk G, Hutchinson P, van der Jagt M, Jain S, Jain S, Jiang JY, Kent H, Kolias A, Kompanje EJO, Lecky F, Lingsma HF, Maegele M, Majdan M, Markowitz A, McCrea M, Meyfroidt G, Mikolic A, Mondello S, Mukherjee P, Nelson D, Nelson LD, Newcombe V, Okonkwo D, Oresic M, Peul W, Pisica D, Polinder S, Ponsford J, Puybasset L, Raj R, Robba C, Roe C, Rosand J, Schueler P, Sharp DJ, Smielewski P, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Temkin N, Tenovuo O, Theadom A, Thomas I, Espin AT, Turgeon AF, Unterberg A, Van Praag D, van Veen E, Verheyden J, Vyvere TV, Wang KKW, Wiegers EJA, Williams WH, Wilson L, Wisniewski SR, Younsi A, Yue JK, Yuh EL, Zeiler FA, Zeldovich M, Zemek R; InTBIR Participants and Investigators. Traumatic brain injury: progress and challenges in prevention, clinical care, and research. Lancet Neurol. 2022 Nov;21(11):1004-1060. doi: 10.1016/S1474-4422(22)00309-X. Epub 2022 Sep 29. PMID 36183712
- [Background] Wu S, Wu B, Liu M, Chen Z, Wang W, Anderson CS, Sandercock P, Wang Y, Huang Y, Cui L, Pu C, Jia J, Zhang T, Liu X, Zhang S, Xie P, Fan D, Ji X, Wong KL, Wang L; China Stroke Study Collaboration. Stroke in China: advances and challenges in epidemiology, prevention, and management. Lancet Neurol. 2019 Apr;18(4):394-405. doi: 10.1016/S1474-4422(18)30500-3. PMID 30878104
- [Background] Multi-Society Task Force on PVS. Medical aspects of the persistent vegetative state (1). N Engl J Med. 1994 May 26;330(21):1499-508. doi: 10.1056/NEJM199405263302107. PMID 7818633
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549
- [Background] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973
- [Background] Denison T, Morrell MJ. Neuromodulation in 2035: The Neurology Future Forecasting Series. Neurology. 2022 Jan 11;98(2):65-72. doi: 10.1212/WNL.0000000000013061. PMID 35263267
- [Background] Petersen EA, Stauss TG, Scowcroft JA, Brooks ES, White JL, Sills SM, Amirdelfan K, Guirguis MN, Xu J, Yu C, Nairizi A, Patterson DG, Tsoulfas KC, Creamer MJ, Galan V, Bundschu RH, Paul CA, Mehta ND, Choi H, Sayed D, Lad SP, DiBenedetto DJ, Sethi KA, Goree JH, Bennett MT, Harrison NJ, Israel AF, Chang P, Wu PW, Gekht G, Argoff CE, Nasr CE, Taylor RS, Subbaroyan J, Gliner BE, Caraway DL, Mekhail NA. Effect of High-frequency (10-kHz) Spinal Cord Stimulation in Patients With Painful Diabetic Neuropathy: A Randomized Clinical Trial. JAMA Neurol. 2021 Jun 1;78(6):687-698. doi: 10.1001/jamaneurol.2021.0538. PMID 33818600
- [Background] Hara S, Andresen H, Solheim O, Carlsen SM, Sundstrom T, Lonne G, Lonne VV, Taraldsen K, Tronvik EA, Oie LR, Gulati AM, Sagberg LM, Jakola AS, Solberg TK, Nygaard OP, Salvesen OO, Gulati S. Effect of Spinal Cord Burst Stimulation vs Placebo Stimulation on Disability in Patients With Chronic Radicular Pain After Lumbar Spine Surgery: A Randomized Clinical Trial. JAMA. 2022 Oct 18;328(15):1506-1514. doi: 10.1001/jama.2022.18231. PMID 36255427
- [Background] Mekhail N, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Pope JE, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, Carlson J, Kim CK, Yang MI, Stauss T, Poree L; Evoke Study Group. Long-term safety and efficacy of closed-loop spinal cord stimulation to treat chronic back and leg pain (Evoke): a double-blind, randomised, controlled trial. Lancet Neurol. 2020 Feb;19(2):123-134. doi: 10.1016/S1474-4422(19)30414-4. Epub 2019 Dec 20. PMID 31870766
- [Background] North RB, Kidd DH, Zahurak M, James CS, Long DM. Spinal cord stimulation for chronic, intractable pain: experience over two decades. Neurosurgery. 1993 Mar;32(3):384-94; discussion 394-5. doi: 10.1227/00006123-199303000-00008. PMID 8455763
- [Background] Funahashi K, Komai N, Ogura M, Kuwata T, Nakai M, Tsuji N. [Effects and indications of spinal cord stimulation on the vegetative syndrome]. No Shinkei Geka. 1989 Oct;17(10):917-23. Japanese. PMID 2812256
- [Background] Kanno T, Morita I, Yamaguchi S, Yokoyama T, Kamei Y, Anil SM, Karagiozov KL. Dorsal column stimulation in persistent vegetative state. Neuromodulation. 2009 Jan;12(1):33-8. doi: 10.1111/j.1525-1403.2009.00185.x. PMID 22151220
- [Background] Piedade GS, Assumpcao de Monaco B, Guest JD, Cordeiro JG. Review of spinal cord stimulation for disorders of consciousness. Curr Opin Neurol. 2023 Dec 1;36(6):507-515. doi: 10.1097/WCO.0000000000001222. Epub 2023 Oct 26. PMID 37889524
- [Background] Kinfe TM, Pintea B, Vatter H. Is Spinal Cord Stimulation Useful and Safe for the Treatment of Chronic Pain of Ischemic Origin? A Review. Clin J Pain. 2016 Jan;32(1):7-13. doi: 10.1097/AJP.0000000000000229. PMID 25760739
- [Background] Giacino JT, Katz DI, Schiff ND, Whyte J, Ashman EJ, Ashwal S, Barbano R, Hammond FM, Laureys S, Ling GSF, Nakase-Richardson R, Seel RT, Yablon S, Getchius TSD, Gronseth GS, Armstrong MJ. Practice guideline update recommendations summary: Disorders of consciousness: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; the American Congress of Rehabilitation Medicine; and the National Institute on Disability, Independent Living, and Rehabilitation Research. Neurology. 2018 Sep 4;91(10):450-460. doi: 10.1212/WNL.0000000000005926. Epub 2018 Aug 8. PMID 30089618
- [Background] Thibaut A, Schiff N, Giacino J, Laureys S, Gosseries O. Therapeutic interventions in patients with prolonged disorders of consciousness. Lancet Neurol. 2019 Jun;18(6):600-614. doi: 10.1016/S1474-4422(19)30031-6. Epub 2019 Apr 16. PMID 31003899